CLINICAL TRIAL: NCT01257347
Title: Uncontrolled Hypertension: The Role of Medication Adherence and Clinical Inertia
Brief Title: Measuring Adherence to Control Hypertension
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ian Kronish, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAI1720; K23HL098359 (NIH)
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Medication adherence; clinical inertia; treatment intensification; quality of care
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concealment (control) (Other): Clinicians in the control arm will not receive any electronically-monitored medication adherence information (collected via MedSignals pillbox) at the 1-month visit and will be expected to manage hypertension according to their usual care.
  Interventions: Device: MedSignals pillbox
- Disclosure (intervention) (Experimental): Disclosure of adherence report to clinician:
  At clinic visits with patients with uncontrolled hypertension, clinicians in the intervention arm were provided with a quantitative summary of their patients' electronic adherence to antihypertensive medications (collected via MedSignals pillbox).
  Interventions: Behavioral: Disclosure of adherence report to clinician; Device: MedSignals pillbox

INTERVENTIONS:
Behavioral: Disclosure of adherence report to clinician — During clinical visits with patients with uncontrolled hypertension, clinicians will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. The summary will be in the form of a report that fits onto one page and lists the percent of days patients correctly adhered to each of the monitored BP medications and the mean adherence to the whole regimen. Adherence data will be provided for the 7-days and 1-month prior to the clinic visit. The report will also show the number of days patients exceeded the recommended number of pill container openings. Clinicians in the intervention arm will get a brief training (<10 minutes) in the interpretation and use of the report at the time of enrollment.
  Arms: Disclosure (intervention)
Device: MedSignals pillbox — (Non-experimental) Patients will be given an electronic pillbox. The device records the date and time when each compartment is opened. Adherence to each BP medication was calculated as the percent of doses taken as prescribed. Patients are informed that their adherence was recorded by the electronic pillbox and might be shared with their clinician depending on randomization.
  Other Names: electronic pillbox

SUMMARY:
The purpose of this study is to test whether accurately measuring patients' adherence to their blood pressure medications with electronic pillbox monitors and then providing clinicians with this information can improve the clinical management of uncontrolled hypertension.

DETAILED DESCRIPTION:
Despite the presence of numerous effective medications, one-half of the adults receiving treatment for hypertension in the United States have uncontrolled blood pressure. At least one-third of these hypertensive patients are not adherent to their blood pressure medications. Given this high rate of non-adherence, clinicians will ideally consider whether their patients are taking their pills before deciding whether to intensify a blood pressure regimen. Yet, in practice, clinicians are often unsure about their patients' level of adherence. This uncertainty limits clinicians' ability to optimally manage hypertension. Electronic medication monitors represent the gold-standard for objectively measuring day-to-day adherence. As a result, they have the potential to best reduce uncertainty regarding medication adherence. The goal of this study is to test whether providing clinicians with an objective measure of medication adherence obtained through electronic monitoring can improve clinician management of uncontrolled hypertension. When data from monitoring indicate poor adherence, it may motivate clinicians to counsel their patients on adherence. Conversely, when data from monitoring indicate good adherence among patients with uncontrolled hypertension, it may motivate clinicians to intensify treatment rather than presume patients were non-adherent.

To test this hypothesis, this study will first enroll and randomize 30 primary care clinicians. Clinicians randomized to the intervention will be trained in the use of a quantitative report that summarizes their patients' adherence to blood pressure medications; they will receive these reports during visits with patients who later get enrolled in the study.

The study will then enroll 300 patients with uncontrolled hypertension from the same clinic. These patients will then have their adherence to up to 4 blood pressure medications measured by an electronic pillbox. The MedSignals® pillbox (LIFETECHniques Inc., San Antonio, TX) is small (5"x3½"x1"), easily portable, and can simultaneous monitor adherence to up to four medications. The device records a pill as taken each time the individual pillbox lid is opened and closed. Data on adherence are easily uploaded (< 1 minute) by connecting the pillbox to a telephone line.

Patients will return to the clinic after 1 month of taking their pills from the electronic pillbox for a visit with a research assistant and their clinician. At this time, data from the pillboxes will be downloaded and used to generate an adherence report. The report will summarize the percent of days that blood pressure medications were taken as prescribed during the monitoring period and will provide guidance on how to take action based on the data. After the report is generated (< 5 minutes), patients will attend visits with their clinicians. Clinicians in the intervention group will receive the adherence report at the time of this visit whereas clinicians in the control group will treat patients according to usual care (without report). Hypertension management during the 1-month clinic visit will be assessed after the visit by 1) reviewing the medical note to determine if clinicians intensified hypertension treatment and 2) surveying patients to determine if clinicians counseled them on adherence. Hypertension management will then be compared between groups.

ELIGIBILITY:
Inclusion criteria

* established diagnosis of hypertension
* prescribed at least one blood pressure (BP) medication
* at least two consecutive clinic visits with elevated BP according to Joint National Committee (JNC-7) guidelines (i.e., BP ≥ 140/90 mmHg or ≥ 130/80 mmHg if diabetes or chronic kidney disease)
* 18 to 80 years old
* at least one prior visit with a clinician enrolled in the study

Exclusion criteria

* severe mental illness
* resided in a long-term care facility
* unable to use the electronic adherence device due to physical or cognitive impairment
* non-English or non-Spanish speaking
* unavailable for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Kronish, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moise N, Davidson KW, Chaplin W, Shea S, Kronish I. Depression and clinical inertia in patients with uncontrolled hypertension. JAMA Intern Med. 2014 May;174(5):818-9. doi: 10.1001/jamainternmed.2014.115. No abstract available. PMID 24615061
- [Background] Kronish IM, Lin JJ, Cohen BE, Voils CI, Edmondson D. Posttraumatic stress disorder and medication nonadherence in patients with uncontrolled hypertension. JAMA Intern Med. 2014 Mar;174(3):468-70. doi: 10.1001/jamainternmed.2013.12881. No abstract available. PMID 24296721
- [Background] Alcantara C, Edmondson D, Moise N, Oyola D, Hiti D, Kronish IM. Anxiety sensitivity and medication nonadherence in patients with uncontrolled hypertension. J Psychosom Res. 2014 Oct;77(4):283-6. doi: 10.1016/j.jpsychores.2014.07.009. Epub 2014 Jul 15. PMID 25280825
- [Background] Moise N, Schwartz J, Bring R, Shimbo D, Kronish IM. Antihypertensive drug class and adherence: an electronic monitoring study. Am J Hypertens. 2015 Jun;28(6):717-21. doi: 10.1093/ajh/hpu199. Epub 2014 Oct 24. PMID 25344354
- [Background] Gallagher BD, Muntner P, Moise N, Lin JJ, Kronish IM. Are two commonly used self-report questionnaires useful for identifying antihypertensive medication nonadherence? J Hypertens. 2015 May;33(5):1108-13. doi: 10.1097/HJH.0000000000000503. PMID 25909704
- [Result] Kronish IM, Moise N, McGinn T, Quan Y, Chaplin W, Gallagher BD, Davidson KW. An Electronic Adherence Measurement Intervention to Reduce Clinical Inertia in the Treatment of Uncontrolled Hypertension: The MATCH Cluster Randomized Clinical Trial. J Gen Intern Med. 2016 Nov;31(11):1294-1300. doi: 10.1007/s11606-016-3757-4. Epub 2016 Jun 2. PMID 27255750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers (the cluster units) and patients were recruited from 2010 to 2014 from 2 hospital-based primary care clinics in New York City.
Pre-assignment Details: 200 patients were consented for the run-in and 100 were eligible for the trial and data analysis. 24 out of 49 primary care providers recruited had patients in the trial.
Groups:
- Usual Care Control: Physicians: Clinicians in the control arm will not receive any electronically-monitored medication adherence information at the 1-month visit and will be expected to manage hypertension according to their usual care.35 patients belonged to providers in the control group.
- Electronically-Measuring Adherence Intervention: Physicians: Electronically-measuring adherence to antihypertensive medications: During clinical visits with patients with uncontrolled hypertension, clinicians in the intervention arm will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. The summary will be in the form of a report that fits onto one page and lists the percent of days patients correctly adhered to each of the monitored BP medications and the mean adherence to the whole regimen. Adherence data will be provided for the 7-days and 1-month prior to the clinic visit. The report will also show the number of days patients exceeded the recommended number of pill container openings, and will list suggested clinical actions according to adherence status. Clinicians in the intervention arm will get a brief training (<10 minutes) in the interpretation and use of the report at the time of enrollment. 65 patients belonged to providers in the intervention group.
- Usual Care Control: Patients: Patients with uncontrolled hypertension - during clinical visits, clinicians will not be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications.
- Electronically-Measuring Adherence Intervention: Patients: Patients with uncontrolled hypertension - during clinical visits, clinicians will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications.
Period: Overall Study
Arm/Group | Usual Care Control: Physicians | Electronically-Measuring Adherence Intervention: Physicians | Usual Care Control: Patients | Electronically-Measuring Adherence Intervention: Patients
Started | 12 (Median patients per provider = 3; range 1-10 (35 patients)) | 12 (Median patients per provider = 4; range 1-13 (65 patients)) | 35 | 65
Completed | 12 | 12 | 35 | 65
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 12 usual care clinicians had visits with 35 patients; 12 intervention clinicians has visits with 65 patients. 'Participant' in this study could mean a clinician or a patient.
Groups:
- Usual Care Control: Physicians: Clinicians in the control arm will not receive any electronically-monitored medication adherence information at the 1-month visit and will be expected to manage hypertension according to their usual care.
- Electronically-measuring Adherence: Electronically-measuring adherence to antihypertensive medications: During clinical visits with patients with uncontrolled hypertension, clinicians in the intervention arm will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. The summary will be in the form of a report that fits onto one page and lists the percent of days patients correctly adhered to each of the monitored BP medications and the mean adherence to the whole regimen. Adherence data will be provided for the 7-days and 1-month prior to the clinic visit. The report will also show the number of days patients exceeded the recommended number of pill container openings, and will list suggested clinical actions according to adherence status. Clinicians in the intervention arm will get a brief training (<10 minutes) in the interpretation and use of the report at the time of enrollment.
- Total: Total of all reporting groups
Arm/Group | Usual Care Control: Physicians | Electronically-measuring Adherence | Usual Care Control: Patients | Electronically-Measuring Adherence Intervention: Patients | Total
Number analyzed (Participants) | 12 | 12 | 35 | 65 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 48 (10) | 64 (9) | 64 (8) | 47 (11)
Sex/Gender, Customized [Number; unit: participants]
  Female | 6 | 7 | 22 | 50 | 13
  Male | 6 | 5 | 13 | 15 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 1 | 28 | 47 | 4
  Not Hispanic or Latino | 9 | 11 | 7 | 18 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 18 | 25 | 1
  White | 10 | 9 | 8 | 17 | 19
  More than one race | 0 | 0 | 2 | 4 | 0
  Unknown or Not Reported | 2 | 2 | 7 | 18 | 4
Region of Enrollment [Number; unit: Participants]
  United States | 12 | 12 | 35 | 65 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Visits With Appropriate Hypertension Management
Description: This is assessed using an algorithm in which patients are categorized as adherent or non-adherent based on electronic monitoring. If patients are adherent (summary measure of adherence to blood pressure medications in the week prior to visit is ≥ 80%), then hypertension management is appropriate if clinicians intensify the hypertension regimen or order testing for secondary hypertension. If patients are non-adherent (summary measure of adherence < 80%), then hypertension management is appropriate if clinicians take action to increase adherence through counseling or regimen simplification.
Time Frame: 1 month clinic visit
Measure: Number; unit: percentage of patient-clinician visits
Groups:
- Usual Care Control Group: Clinicians in the control arm will not receive any electronically-monitored medication adherence information at the 1-month visit and will be expected to manage hypertension according to their usual care.
- Electronically-measuring Adherence: At clinical visits with patients with uncontrolled hypertension, clinicians in the intervention arm will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. The summary will be in the form of a report that fits onto one page and lists the percent of days patients correctly adhered to each of the monitored BP medications and the mean adherence to the whole regimen. Adherence data will be provided for the 7-days and 1-month prior to the clinic visit. The report will also show the number of days patients exceeded the recommended number of pill container openings. The report will also provide suggested clinical actions according to adherence status. Clinicians in the intervention arm will get a brief training (<10 minutes) in the interpretation and use of the report at the time of enrollment.
Arm/Group | Usual Care Control Group | Electronically-measuring Adherence
Number analyzed (Participants) | 35 | 65
percentage of patient-clinician visits | 34 | 69
Statistical Analysis 1: Comparison: Usual Care Control Group vs Electronically-measuring Adherence; The sample size was calculated to have sufficient power to detect meaningful differences in appropriateness of clinician management between intervention and control groups. Each patient-clinician encounter was treated as independent and the sample size was inflated to account for the design effect (DE) of clustering of patients within clinician. GEE stands for generalized estimating equation; Test type: Superiority or Other; p <= 0.001, GEE model — We included a stopping rule in which recruitment would be stopped at the midpoint for futility if the z-score was negative or for efficacy if the z-score was positive and the p-value ≤ 0.001; GEE models (logit link) with clinician as the cluster variable, appropriateness of management as outcome, intervention group as explanatory variable

2. Secondary Outcome: Percentage of Visits With Regimen Intensification During 1-month Visit, Adherent in Week Prior to Outcome Visit, Only
Description: This will be determined based on abstracting information from the electronic medical record after the 1-month visit using a standardized instrument. An outcome assessor who is blinded to clinician and patient group assignment will assess whether, during the 1-month visit, the provider intensified the blood pressure regimen (added or increased dose of medications). All prescribing and test ordering at the recruitment clinic is recorded in the electronic medical record.
Time Frame: 1 month clinic visit
Measure: Number; unit: percentage of patient-clinician visits
Groups:
- Usual Care Control Group, Adherent Only: At clinical visits with patients with uncontrolled hypertension, clinicians will not be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. Clinicians will be expected to manage hypertension according to usual care.
- Electronically-measuring Adherence Group, Adherent Only: At clinical visits with patients with uncontrolled hypertension, clinicians in the intervention arm will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. The summary will be in the form of a report that fits onto one page and lists the percent of days patients correctly adhered to each of the monitored BP medications and the mean adherence to the whole regimen. Adherence data will be provided for the 7-days and 1-month prior to the clinic visit. The report will also show the number of days patients exceeded the recommended number of pill container openings. The report will also provide suggested clinical actions according to adherence status. Clinicians in the intervention arm will get a brief training (<10 minutes) in the interpretation and use of the report at the time of enrollment.
Arm/Group | Usual Care Control Group, Adherent Only | Electronically-measuring Adherence Group, Adherent Only
Number analyzed (Participants) | 19 | 34
percentage of patient-clinician visits | 26 | 56

3. Secondary Outcome: Percentage of Visits With Counseling Performed During 1-month Visit, Non-adherent in Week Prior to Outcome Visit or Over Entire Monitoring Period
Description: This will be determined based on interviewing patients immediately after the 1-month visit using a standardized questionnaire. A research assistant who is blinded to group assignment will ask patients questions that assess whether clinicians counseled them about taking their blood pressure medications during that most recent visit. These questions are adapted from a validated questionnaire that assesses provider communication about blood pressure medications.
Time Frame: 1 month clinic visit
Measure: Number; unit: percentage of patient-clinician visits
Groups:
- Usual Care Control Group, Non-adherent Only: Clinicians in the control arm will not receive any electronically-monitored medication adherence information at the 1-month visit and will be expected to manage hypertension according to their usual care.
- Electronically-measuring Adherence Group, Non-adherent Only: At clinical visits with patients with uncontrolled hypertension, clinicians in the intervention arm will be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. The summary will be in the form of a report that fits onto one page and lists the percent of days patients correctly adhered to each of the monitored BP medications and the mean adherence to the whole regimen. Adherence data will be provided for the 7-days and 1-month prior to the clinic visit. The report will also show the number of days patients exceeded the recommended number of pill container openings. The report will also provide suggested clinical actions according to adherence status. Clinicians in the intervention arm will get a brief training (<10 minutes) in the interpretation and use of the report at the time of enrollment.
Arm/Group | Usual Care Control Group, Non-adherent Only | Electronically-measuring Adherence Group, Non-adherent Only
Number analyzed (Participants) | 18 | 32
percentage of patient-clinician visits | 39 | 84

4. Secondary Outcome: Percentage of Visits With Hypertension Regimen Simplification, Non-adherent in Week Prior to Outcome Visit or Over Entire Monitoring Period
Description: This will be determined by abstracting data from the electronic medical record after the 1-month visit using a standardized instrument. An outcome assessor who is blinded to clinician and patient group assignment will assess whether, during the 1-month visit, the provider simplified the regimen by switching from a short-acting, multi-day dosing medication to a long-acting, once per day medication or switched two medication to a single combination pill. All prescribing and test ordering at the recruitment clinic is recorded in the electronic medical record.
Time Frame: 1 month clinic visit
Population: patient-provider visits
Measure: Number; unit: percentage of patient-clinician visits
Groups:
- Usual Care Control Group, Non-adherent Only: At clinical visits with patients with uncontrolled hypertension, clinicians will not be provided with a quantitative summary of their patients' electronically-monitored adherence to antihypertensive medications. Clinicians will be expected to manage hypertension according to usual care.
Arm/Group | Usual Care Control Group, Non-adherent Only | Electronically-measuring Adherence Group, Non-adherent Only
Number analyzed (Participants) | 18 | 32
percentage of patient-clinician visits | 6 | 9

ADVERSE EVENTS:
Time Frame: Interval between enrollment visit and next scheduled primary care visit (mean 52 days, standard deviation 32 days).
Groups:
- Usual Care Control: Physicians: Clinicians in the control arm will not receive any electronically-monitored medication adherence information at the 1-month visit and will be expected to manage hypertension according to their usual care. 35 patients belonged to providers in the control group.
Arm/Group | Usual Care Control: Physicians | Electronically-Measuring Adherence Intervention: Physicians | Usual Care Control: Patients | Electronically-Measuring Adherence Intervention: Patients
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/35 | 0/65
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/35 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No